CLINICAL TRIAL: NCT01635296
Title: A Multicenter, Open Label, Phase 1B Study of Escalating Doses of RO5045337 Administered Orally, With Cytarabine Administered A) Subcutaneously, or B) Intravenously, in Patients With Acute Myelogenous Leukemia (AML)
Brief Title: A Study of RO5045337 in Combination With Cytarabine in Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28023; 2011-006252-36 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-07-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Myelogenous Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

ARMS (2):
- A: Previously untreated (Experimental)
  Interventions: Drug: RO5045377; Drug: cytarabine
- B: Relapse/Refractory (Experimental)
  Interventions: Drug: RO5045377; Drug: cytarabine

INTERVENTIONS:
Drug: RO5045377 — Multiple escalating oral doses, Days 1 to 10 of each 28-day cycle
  Arms: A: Previously untreated
Drug: RO5045377 — Multiple escalating oral doses, Days 1 to 5 of each 28-day cycle
  Arms: B: Relapse/Refractory
Drug: cytarabine — 20 mg/m2 sc, Days 1 to 10 of each 28-day cycle
  Arms: A: Previously untreated
Drug: cytarabine — 1 gm/m2 iv, Days 1 to 6 of each 28-day cycle
  Arms: B: Relapse/Refractory

SUMMARY:
This multi-center, open-label, Phase 1b study will evaluate the safety, pharmacokinetics and efficacy of RO5045337 in combination with cytarabine in patients with acute myelogenous leukemia. In Arm A, cohorts of previously untreated patients deemed unsuitable for standard induction therapy will receive escalating oral doses of RO5045377 and cytarabine 20 mg/m2 subcutaneously daily for Days 1 to 10 of each 28-day cycle. In Arm B, cohorts of patients who have relapsed or are refractory after at least one cytarabine/anthracycline containing regimen will receive escalating oral doses of RO5045377 on Days 1 to 5 and cytarabine 1 gm/m2 intravenously on Days 1 to 6 of each 28-day cycle. Patients will receive up to 4 cycles of therapy, patients in Arm A who achieve hematologic response may continue additional cycles until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with histologically or cytologically documented acute myelogenous leukemia appropriate for cytarabine therapy including:
* Arm A: Patients who have not received prior standard induction chemotherapy, considered unsuitable for standard induction therapy
* Arm B: Patients who have failed their 1st or greater line of standard induction chemotherapy (primary refractory) or patients who originally achieved a complete response but are currently in first or greater relapse
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* All non-hematological adverse events of any prior chemotherapy, surgery, or radiotherapy must have resolved to NCI-CTC AE Grade </=2
* Adequate hepatic and renal function
* Patient must be willing to submit the blood sampling and bone marrow sampling for PK and PD analyses and exploratory biomarkers

Exclusion Criteria:

* History of allergic or toxic reactions attributed to cytarabine or a history of allergic reactions to components of the formulated product
* Current evidence of CNS leukemia
* Any severe and/or uncontrolled medical condition or other conditions that could affect the participation in the study
* Pregnant or breastfeeding women
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose/dose-limiting toxicities | approximately 12 months
Safety: Incidence of adverse events | approximately 12 months

SECONDARY OUTCOMES:
Efficacy: Hematologic response | approximately 1 year
Pharmacodynamics: Biomarkers (MIC-1, protein, nucleic acid, other) from bone marrow/buccal tissue/blood | Pre-dose (and up to 12 hours post-dose Day 1 and Day 10 or Day 5)
Pharmacokinetics: Cmax/area under the concentration-time curve | Pre-dose and up to 12 hours post-dose Day 1 and Day 10 or Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (3):
  - Valhalla, New York
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Marseille, France
- Bologna, Emilia-Romagna, Italy
- United Kingdom (2):
  - Glasgow
  - Manchester